CLINICAL TRIAL: NCT04228341
Title: The Effect of Degree of Rice-polishing on Glycaemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/01079
Record Dates: First submitted 2020-01-11; First posted 2020-01-14 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Glucose Reference 1 (Other): Glucose solution 1
  Interventions: Other: Glucose Reference 1
- Glucose Reference 2 (Other): Glucose solution 2
  Interventions: Other: Glucose Reference 2
- Glucose Reference 3 (Other): Glucose solution 3
  Interventions: Other: Glucose Reference 3
- Brown Rice (Experimental): Cooked brown rice
  Interventions: Other: Brown Rice
- 3 % polished rice (Experimental): Cooked 3 % polished rice
  Interventions: Other: 3 % polished rice
- 6 % polished rice (Experimental): Cooked 6 % polished rice
  Interventions: Other: 6 % polished rice
- 9 % polished rice (Experimental): 9 % polished rice
  Interventions: Other: 9 % polished rice
- 20 % Polished rice (Experimental): Cooked 20 % Polished rice (White Rice)
  Interventions: Other: 20 % Polished rice

INTERVENTIONS:
Other: Glucose Reference 1 — 50 g of glucose dissolved in 250 ml of water (First glucose control visit)
  Arms: Glucose Reference 1
Other: Glucose Reference 2 — 50 g of glucose dissolved in 250 ml of water (Second glucose control visit)
  Arms: Glucose Reference 2
Other: Glucose Reference 3 — 50 g of glucose dissolved in 250 ml of water (Third glucose control visit)
  Arms: Glucose Reference 3
Other: Brown Rice — Unpolished brown rice containing 50 g of available carbohydrate was cooked using a rice cooker (Toyomi) at a ratio of rice to water of 1: 2
  Arms: Brown Rice
Other: 3 % polished rice — 3% polished rice, containing 50 g of available carbohydrate was cooked using a rice cooker at a ratio of rice to water of 1: 2
  Arms: 3 % polished rice
Other: 6 % polished rice — 6% polished rice, containing 50 g of available carbohydrate was cooked using a rice cooker at a ratio of rice to water of 1: 2
  Arms: 6 % polished rice
Other: 9 % polished rice — 9 % polished rice, containing 50 g of available carbohydrate was cooked using a rice cooker at a ratio of rice to water of 1: 2
  Arms: 9 % polished rice
Other: 20 % Polished rice — White rice (20% polished rice), containing 50 g of available carbohydrate was cooked using a rice cooker at a ratio of rice to water of 1: 2.
  Arms: 20 % Polished rice

SUMMARY:
To investigate the effects of rice polishing on glycaemic and insulinaemic response in healthy Chinese male volunteers.

DETAILED DESCRIPTION:
There will be a total of 8 test session. Each session will last for 3.5 hours. At each test session, volunteers will be served with test meal and blood will be collected. After an overnight fast, subjects will visit the research center. Two fasting capillary blood samples will be collected via fingerprick. Following the fasting samples, subject will consume the test meals. Further blood samples will be collected at 15, 30, 45, 60, 90, 120, 150, 180 minutes after the ingestion of test meal. These samples will be used to analyses for whole capillary blood glucose. At every 30 minute interval, samples will be collected for analysis of capillary plasma insulin.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese ethnicity
* Age ≥21 and ≤ 60 years
* Body mass index between 18.5 to 25 kg/m2
* Normal blood pressure =<140/90 mmHg
* Fasting blood glucose <6.0 mmol/L
* In general good health

Exclusion Criteria:

* Current smoker
* Have any metabolic diseases (such as diabetes, hypertension etc)
* Do not have known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Have medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Have intolerances or allergies to any foods
* Currently partake in sports at the competitive and/or endurance levels
* Intentionally restrict food intake

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male only
Enrollment: 14 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Glucose | Up to 180 minutes
  Whole capillary blood glucose will be measure using Hemocue analyser

SECONDARY OUTCOMES:
Insulin | Up to 180 minutes
  Capillary plasma will be measure using Cobas analyser

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No